CLINICAL TRIAL: NCT05497154
Title: Physical Therapists Identifying Patients With Opioid Misuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jake Magel, Research Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3394
Record Dates: First submitted 2022-08-03; First posted 2022-08-11 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Opioid Misuse; Musculoskeletal Pain
Keywords: opioid misuse; physical therapy; physical therapist
MeSH Terms: conditions — Opioid-Related Disorders; Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training Arm (Experimental)
  Interventions: Behavioral: Training Arm

INTERVENTIONS:
Behavioral: Training Arm — The training will be composed of 4 separate training sessions provided every 2 - 4 weeks. During the 1st session (45 minutes), the investigators will educate the physical therapist about the different categories of opioid use including opioid misuse (OM) and the risks associated with OM as well as training to engage the patient in a conversation about opioid use. The 2nd and 3rd sessions (30 minutes each) involve training in procedures to screen and assess patients at risk for OM, respectively. The 4th session (30 minutes) involves training in procedures to refer patients to a specialist or a primary care provider for further treatment if OM is suspected.

SUMMARY:
The purpose of this study is to develop and operationalize key procedures for physical therapists (n = 12) to address patients who are at risk for or have opioid misuse (OM). The investigators will train physical therapists in procedures to: 1) engage patients at risk for OM in conversations about appropriate opioid use, 2) screen and 3) assess these patients for OM and, 4) refer patients for further treatment if OM is suspected. The investigators will employ a modified Delphi approach to iteratively refine and operationalize the procedures and to arrive at a finalized procedure manual followed by an evaluation of the implementation of these procedures.

DETAILED DESCRIPTION:
The purpose of this study is to develop and operationalize key procedures for physical therapists (n = 12) to address patients who are at risk for or have OM. The investigators will train physical therapists in procedures to: 1) engage patients at risk for OM in conversations about appropriate opioid use, 2) screen and 3) assess these patients for OM and, 4) refer patients for further treatment if OM is suspected. The investigators will employ a modified Delphi approach to iteratively refine and operationalize the procedures and to arrive at a finalized procedure manual followed by an evaluation of the implementation of these procedures. Approximately 4 months following the development of the manual and the distribution of the finalized manual, the investigators will conduct semi-structured interviews to determine the barriers and facilitators to implementing the procedures learned in the training.

Our aims are:

1. Qualitatively evaluate physical therapists' perceptions and recommendations for implementing OM procedures.
2. Evaluate the implementation of the manualized OM procedures.

ELIGIBILITY:
Inclusion Criteria:

* University of Utah physical therapists with at least 0.5 full-time equivalent
* Self report managing patients with musculoskeletal pain

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-05-27 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Change in the Drug and Drug Problems Perception Questionnaire (DDPPQ) | Baseline, immediate post training, 4 months after last training session
  The DDPPQ is a 20 item tool used to measure the attitudes of health care providers related to the management of patients misusing drugs and contains 5 subscales (Role Adequacy: 7 items; Role Legitimacy: 2 items; Role Support: 3 items; Role Self-esteem: 4 items; Job Satisfaction: 4 items) Each item is scored on a 7-point scale (1 = strongly agree to 7 = strongly disagree). Each item was modified to asses the health care providers' attitudes about managing patients with opioid misuse.

OTHER OUTCOMES:
Thematic analysis from semi-structured interviews | 4 months after the last training session
  Semi-structured interviews to assess barriers and facilitators of implementing the procedures learned in the training
Reach | Immediate post training
  Proportion of physical therapists who agreed to attend the training that attended all training sessions
Adoption 1- engaging patients in conversations | Approximately 4 months after last training session
  Percentage of physical therapists who attended the training that report engaging patients in conversations about opioid misuse,
Adoption 2 - screening | Approximately 4 months after last training session
  Percentage of physical therapists who attended the training that report screening for opioid misuse
Adoption 3 - assessing | Approximately 4 months after last training session
  Percentage of physical therapists who attended the training that report assessing patients for opioid misuse
Adoption 4 - referring | Approximately 4 months after last training session
  Percentage of physical therapists who attended the training that report referring for opioid misuse
Qualitative thematic analysis of each focus group | Immediately after each of the 4 training sessions.
  The investigators will conduct focus groups after each training session. All sessions will be analyzed together to qualitatively assess the physical therapists' receptivity to the procedures learned in the training sessions.
Change in the Frequency of opioid misuse management practices - Adapted from the Alcohol Education Survey | Baseline, immediately post training and to approximately 4 months after the last training session
  Questions were adapted: "How often do you ask patients about alcohol problems?" was modified to: "How often do you ask patients about problems with prescription opioid medication misuse? 4 additional questions were similarly modified ([1] How often do you formally screen patients for prescription opioid medication misuse using screening instruments, such as the Current Opioid Misuse Measure or other tools; [2] How often do you assess patients' readiness to change their prescription opioid medication misuse behaviors?; [3] How often do you discuss/advise patients to change their prescription opioid medication misuse behaviors?; [4] How often do you refer patients with prescription opioid medication misuse for further assessments or interventions?). Scoring: Never, Rarely (less than 10% of the time), Occasionally (about 30% of the time), Sometimes (about 50% of the time), Frequently (about 70% of the time), Usually (about 90% of the time), Every time.
Manual of procedures | Approximately 4 months after the last training session.
  At the end of the study after the individual interviews, the investigators will finalize the manual of opioid misuse procedures for physical therapists.
Change in the Confidence in opioid misuse management practices. Adapted from the Alcohol Education Survey | Baseline, immediately post training and to approximately 4 months after the last training session
  These questions were adapted from a survey developed to improve health care providers' management of patients with alcohol problems. The questions are: ([1] I am confident in my ability to ask patients about prescription opioid medication misuse, [2] I am confident in my ability to formally screen patients for prescription opioid medication misuse using screening instruments, such as the Current Opioid Misuse Measure or other tools; [3] I am confident in my ability to assess patients' readiness to change their prescription opioid medication misuse behaviors; [4] I am confident in my ability to discuss/advise patients to change their prescription opioid medication misuse behaviors; [5] I am confident in my ability to refer patients with prescription opioid medication misuse for further assessments or interventions?). Each confidence with management practice question was scored on a 7-point Likert scale (1 = no confidence; 7 = high confidence).

CONTACTS AND LOCATIONS:
Overall Officials: John Magel, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared: Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
  What documents will be available: Study protocol, statistical analysis plan, Analytic code.
  With whom will the data be shared: Researchers who provide a methodologically sound proposal
  For what type of analyses: To achieve the aims in approved proposal
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: By what mechanism will data be made available: Proposal should be directed to Jake.Magel@hsc.utah.edu to gain access, data requestors will need to sign a data access agreement. Link to data will be provided.

REFERENCES:
- [Background] D'Onofrio G, Nadel ES, Degutis LC, Sullivan LM, Casper K, Bernstein E, Samet JH. Improving emergency medicine residents' approach to patients with alcohol problems: a controlled educational trial. Ann Emerg Med. 2002 Jul;40(1):50-62. doi: 10.1067/mem.2002.123693. PMID 12085073
- [Background] Watson H, Maclaren W, Kerr S. Staff attitudes towards working with drug users: development of the Drug Problems Perceptions Questionnaire. Addiction. 2007 Feb;102(2):206-15. doi: 10.1111/j.1360-0443.2006.01686.x. PMID 17222274